CLINICAL TRIAL: NCT01418976
Title: IMPROVING WALKING AND BALANCE IN VETERANS WITH TRAUMATIC BRAIN INJURY: A PILOT STUDY EXAMINING FEASIBILITY AND DOSAGE
Brief Title: Walking and Balance Post-TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: INTRuST, Post-Traumatic Stress Disorder - Traumatic Brain Injury Clinical Consortium (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INTRuST-Walking and Balance; Pro00007596 (Other: University of South Carolina IRB)
Record Dates: First submitted 2011-08-16; First posted 2011-08-17 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Difficulties, Ambulation; Brain Injuries, Traumatic
Keywords: physical therapy techniques; brain injuries, traumatic; walking; gait; postural balance
MeSH Terms: conditions — Mobility Limitation; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intensive Mobility Training (IMT) (Experimental): Intensive Mobility Training will be used as an intensive physical therapy intervention. Participants will receive 3 hours per day for a 10 day session, be post-tested, and receive another 10 day session followed by two more testing sessions.
  Interventions: Behavioral: Intensive Mobility Training (IMT)

INTERVENTIONS:
Behavioral: Intensive Mobility Training (IMT) — Intensive Mobility Training will be used as an intensive physical therapy intervention. Participants will receive 3 hours per day for a 10 day session, be post-tested, and receive another 10 day session followed by two more testing sessions.

SUMMARY:
This is a case series study evaluating the feasibility and dosage of Intensive Mobility Training (IMT). Twelve participants with chronic, mild-to-moderate, Traumatic Brain Injury (TBI) causing significant locomotor impairment, who meet these specific criteria, will be recruited. Location and nature of neural insult will be determined by multimodal Magnetic Resonance Imaging (MRI) exam. All participants will receive 3 hours of rehabilitation per day for 20 days, focusing on gait and balance. Locomotion and balance will be comprehensively tested prior to IMT, after 10 days of IMT, and then again after the full dose of IMT. This study will determine the feasibility of this intervention in the population of TBI patients, allow an estimate of effect size and provide initial information on possible neural predictors of success. Furthermore the investigators will be able to determine whether the dosage of 10 days is sufficient or whether significant improvements are made with 20 days of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. greater than 3 months post-TBI (as defined by INTRuST criteria) and no longer receiving care as an inpatient in a rehabilitation facility.
2. the ability to follow simple three-step commands;
3. the ability to communicate presence and location of pain;
4. the ability to sit independently without back or arm support for five minutes;
5. the ability to stand with support of a straight cane, quad cane, or walker for 2 minutes;
6. the ability to walk 10 meters with maximum 1 person assisting;
7. presence of motor deficits (determined by clinical assessment of paresis);
8. age ≥ 18;
9. ability to give consent or have a acceptable surrogate capable of giving consent on subject's behalf

Exclusion Criteria:

1. unable to ambulate 500 feet prior to TBI;
2. history of serious chronic obstructive pulmonary disease or oxygen dependence;
3. severe weight bearing pain;
4. lower-extremity amputation;
5. non-healing ulcers on the lower-extremity;
6. renal dialysis or end stage liver disease;
7. legal blindness or severe visual impairment;
8. severe arthritis or orthopedic problems that limit passive ranges of motion of lower extremity (knee flexion contracture of -10°, knee flexion Range of Motion < 90°, hip flexion contracture > 25°, and ankle plantar flexion contracture > 15°);
9. history of deep venous thrombosis or pulmonary embolism within 6 months
10. uncontrollable diabetes with recent weight loss, diabetic coma, or frequent insulin reactions;
11. severe hypertension with systolic greater than 200 mmHg and diastolic greater than 110 mmHg at rest;
12. intracranial hemorrhage related to aneurysm rupture or an arteriovenous malformation (hemorrhagic infarctions will not be excluded);
13. history of severe uncontrolled seizure disorder;
14. other neurological conditions such as multiple sclerosis or Parkinson's Disease;
15. pain that is scored greater than 5 out of 10 on a visual analog scale;
16. any factor contraindicative to MRI examination (e.g., cardiac pacemaker/ defibrillator, pregnancy, aneurysm clips, insulin pump, metal fragments in the body).
17. any other health problems judged by their screening physician to put the client at significant risk of harm during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Feasibility as measured by study completion. | post-treatment (after 20-day intervention)
  Feasibility will be determined by the ratio of participants that complete the intervention.
Feasibility as measured by pain ratings. | during 20-day intervention
  Feasibility will be determined by daily change in pain scores as measured using visual analog scales.
Feasibility as measured by fatigue ratings. | during 20-day intervention
  Feasibility will be determined by daily change in fatigue scores as measured using visual analog scales.

SECONDARY OUTCOMES:
Efficacy as measured by improvements in gait and mobility. | from pre- to post-treatment during 20-day intervention.
  Efficacy will be measured by improvements in mobility and gait as measured by the Dynamic Gait Index, Timed Up and Go, Six- Minute Walk, and Falls Efficacy Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Fritz, Ph.D., P.T., Principal Investigator — University of South Carolina
Locations (1):
- 921 Assembly Street, 3rd Floor, Public Health Research Center, University of South Carolina, Columbia, South Carolina, United States